CLINICAL TRIAL: NCT01848444
Title: Evaluation of Different Chemical Substances in the Milk of Breastfed Infant
Brief Title: Levels of Contaminants in Human Milk
Acronym: Conta-Lait
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 12009; CRC12014 (Other: Assistance publique)
Record Dates: First submitted 2013-04-18; First posted 2013-05-07 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Lactating Women Who Give Their Milk to One of the 6 Milk Banks Participating in the Study
Keywords: Public Health; Epidemiology; Pharmacy Toxicology; Perinatal period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4*200 ml of breastmilk homogenizated and frozen -18° Celsius in the milk bank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lactating women who give her breastmilk to a milkbank: 180 women will be included in 6 milk banks in France during 18 months
  Interventions: Other: Breastmilk

INTERVENTIONS:
Other: Breastmilk — to measure levels of contaminants in human breastmilk samples

SUMMARY:
Recent international data have shown that the levels of chemical substances found in human milk could be at risk for breastfed infants. New data are necessary to assess this risk among French newborns.

DETAILED DESCRIPTION:
The objective of this study is to assess levels of certain contaminants in breastmilk. Measurements will be made on breastmilk samples collected in Milk Bank but not suitable for infants due to bacteriological reasons. 6 Milk Banks well distributed on the French territory will be contacted to participate. 180 women will be included. Women who gave their milk and correspond to the inclusion criteria (in particular breastfeeding a child under 6 months at the time of the donation) will be contacted by the investigator by phone. They will be asked to fill in a written consent as well as a questionnaire on socio-demographic data, pregnancy related information and potential environmental exposures.

2 breastmilk samples of 50 mL will be sendsending to the lab for analysis and 2 samples of 50 mL will be collected.

ELIGIBILITY:
Inclusion Criteria:

For the samples:

* Not allowed to use for bacteriological reasons
* Breastmilk samples from lactating women between delivery and 6 months (+/- 1 month) of the infant

For the mothers:

* Age > or = 18 years
* Lived on the French territory
* Well french writer and speaker
* Mother child couple in good health
* Non opposability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lactating women given their milk to a milk bank
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Presence of contaminants (PCB, dioxins, furans and brominated flame retardants) | at the moment of the milk's donation
  analysis of contaminants

SECONDARY OUTCOMES:
evaluate the concentration of other contaminants, perfluorinated compounds, organochlorine pesticides and inorganic compounds | at the moment of the milk's donation
  analysis of contaminants
To estimate the exposure of breastfed infants and to assess the risk in this population | at the moment of the milk's donation
  statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Rigourd, MD, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Hopital Necker, Paris, France